CLINICAL TRIAL: NCT02898753
Title: A Three-Month, Open-Label, Randomized, Dose-escalation Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of VAL-1221 Versus Myozyme®/Lumizyme® in Patients With Late-Onset GSD-II (Pompe Disease) Followed by Open-Label Treatment With VAL-1221 in All Patients
Brief Title: VAL-1221 Delivered Intravenously in Ambulatory and Ventilator-free Participants With Late-Onset Pompe Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company closure due to lack of funding
Sponsor: Valerion Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAL1221-201-16
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Pompe Disease
Keywords: GSD-II; Pompe Disease; Glycogen Storage Diseases; GAA
MeSH Terms: conditions — Glycogen Storage Disease Type II; Glycogen Storage Disease | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VAL-1221 3 mg/kg (Experimental): Part 1: Participants will receive VAL-1221 3 mg/kg IV infusion every other week for 12 weeks, inclusive, for a total of 7 infusions.
  Part 2: Participants from Part 1 of the study who were randomized to VAL-1221 3 mg/kg can enter Part 2 of the study and receive VAL-1221 at a dose of 3 mg/kg IV infusion every other week. The dose can be increased by the Investigator to 10 mg/kg and further to 30 mg/kg (after at least 12 weeks of dosing at 10 mg/kg), depending upon the pharmacodynamics, efficacy, and safety data.
  Interventions: Drug: VAL-1221
- VAL-1221 10 mg/kg (Experimental): Part 1: Participants will receive VAL-1221 10 mg/kg IV infusion every other week for 12 weeks, inclusive, for a total of 7 infusions.
  Part 2: Participants from Part 1 of the study who were randomized to VAL-1221 10 mg/kg can enter Part 2 of the study and receive VAL-1221 at a dose of 10 mg/kg IV infusion every other week. The dose can be increased by the Investigator to 30 mg/kg IV infusion, depending upon the pharmacodynamics, efficacy, and safety data.
  Interventions: Drug: VAL-1221
- VAL-1221 30 mg/kg (Experimental): Part 1: Participants will receive VAL-1221 30 mg/kg IV every other week for 12 weeks, inclusive, for a total of 7 infusions.
  Part 2: Participants from Part 1 of the study who were randomized to VAL-1221 30 mg/kg can enter Part 2 of the study and receive VAL-1221 at a dose of 30 mg/kg IV inufsion every other week.
  Interventions: Drug: VAL-1221
- rhGAA (Active Comparator): Part 1: Participants will be maintained on their current dose and regimen of Myozyme or Lumizyme.
  Part 2: Participants from Part 1 of the study who were randomized to rhGAA can enter Part 2 of the study and receive VAL-1221 either 3 mg/kg, 10 mg/kg, or 30 mg/kg (based on the dose of VAL-1221 in respective cohorts to which they were randomized in Part 1) IV infusion every other week.
  Interventions: Drug: VAL-1221; Drug: RhGAA

INTERVENTIONS:
Drug: VAL-1221 — VAL-1221 3, 10, or 30 mg/kg as per the dose and schedule specified in the arm group description
Drug: RhGAA — Active comparator
  Other Names: Myozyme; Lumizyme
  Arms: rhGAA

SUMMARY:
This Phase I/II open-label, randomized, dose-escalation study will assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of VAL-1221 versus Myozyme®/Lumizyme® in participants with late-onset glycogen storage disease-II (GSD-II) (Pompe disease)

DETAILED DESCRIPTION:
Part 1 comprises 3 sequential cohorts of 4 patients each randomized to treatment with either VAL-1221 (at 3, 10, or 30 mg/kg) or positive control (rhGAA). Patients randomized to VAL-1221 will receive 7 intravenous (IV) infusions of VAL-1221 (one infusion every other week) over 12 weeks. Control patients will continue receiving their accustomed dose and regimen of Myozyme®. Part 2 is an uncontrolled extension to evaluate long-term effects of VAL-1221 given by IV infusion once every other week at doses up to 40 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able and willing to provide informed consent prior to any study procedures are performed
* Diagnosis of GSDII based on one of the following:

  * Endogenous cultured skin fibroblast GAA activity less than (<) 40 percent (%) of adult normal level
  * Endogenous whole blood or dried blood spot GAA activity in deficiency range
  * Genetic analysis showing pathogenic variants in both alleles
* Onset of Pompe disease-related symptoms after 1 year of age
* Previously treated with Myozyme or Lumizyme for at least 12 months and on a stable regimen for the past 6 months
* Sexually active participants who are willing to use an acceptable method of contraception (abstinence, oral contraceptives, barrier method with spermicide, surgical sterilization, implanted or injectable contraceptives with a stable dose for at least 1 month prior to Baseline, hormonal intra-uterine device [IUD] inserted at least 1 month prior to Baseline) during the study and for 30 days after completion of treatment

  * If participant is female and not considered to be of childbearing potential, she is at least 2 years post-menopause, has undergone a tubal ligation, a total hysterectomy or bilateral oophorectomy
  * If participant is female and of childbearing potential, she has a negative serum pregnancy test during screening and Baseline and must be willing to undergo pregnancy testing at specific intervals during the study
* Participant meets at least one of the following criteria: greater than (>) 30% and <80% predicted upright forced volume capacity (FVC) or participant is able to walk >20% but <80% predicted normal on 6-minute walk test with or without use of assistive devices
* Able to comply with protocol requirements

Exclusion Criteria:

* Cardiac involvement in first year of life
* Anti-GAA antibody titers >1:51,200 at two time points
* Prior use of chaperone therapy for GSD-II within the last 12 months
* Use of immunosuppressive medication other than glucocorticoids within 6 months prior to study enrollment
* Use of invasive ventilatory assistance other than Bilevel Positive Airway Pressure (BiPAP) at night or during periods of rest
* Has received any investigational medication or has enrolled in any study involving investigational drugs or therapies within 30 days prior to first dose of study drug
* Start of or change in usual regimen of albuterol or respiratory muscle training within 30 days prior to first dose of study drug
* History of sensitivity to any of the constituents of the study drug
* Participant is breastfeeding or planning to become pregnant or to breastfeed during the study or is currently breastfeeding
* Participant has a medical condition or circumstance that, in the opinion of the investigator, might compromise the participant's ability to comply with the protocol or the participant's well-being or safety
* Participant has any condition that, in the view of the investigator, places the participant at high risk of poor treatment compliance or of not completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-related Treatment-emergent Adverse Events (TEAEs) | Baseline of Study Part 1 though Month 24 of Study Part 2
Number of Participants With Infusion-Associated Reactions to VAL-1221 | Baseline of Study Part 1 though Month 24 of Study Part 2
Percentage of Participants with Anti-VAL-1221 Antibodies | Baseline of Study Part 1 though Month 24 of Study Part 2
Percentage of Participants with GAA Antibodies | Baseline of Study Part 1 though Month 24 of Study Part 2

SECONDARY OUTCOMES:
Pharmacokinetics of VAL-1221 in Plasma: Maximum Observed Concentration (Cmax) | Part 1: Pre-infusion, end of infusion (EOI) (infusion duration 1 mg/kg/hour), at 0.25, 0.5, 1, 2, 4, 12, 24, 48 and 336 hours after EOI on Days 1, 2, 3 and Week 12; Part 2: Pre-infusion on Weeks 12, 14, 16, 18, 20, 22, Months 12, 24, 36
Pharmacokinetics of VAL-1221 in Plasma: Time to Reach Maximum Concentration (Tmax) | Part 1: Pre-infusion, end of infusion (EOI) (infusion duration 1 mg/kg/hour), at 0.25, 0.5, 1, 2, 4, 12, 24, 48 and 336 hours after EOI on Days 1, 2, 3 and Week 12; Part 2: Pre-infusion on Weeks 12, 14, 16, 18, 20, 22, Months 12, 24, 36
Pharmacokinetics of VAL-1221 in Plasma: Area Under the Concentration Time Curve (AUC) | Part 1: Pre-infusion, end of infusion (EOI) (infusion duration 1 mg/kg/hour), at 0.25, 0.5, 1, 2, 4, 12, 24, 48 and 336 hours after EOI on Days 1, 2, 3 and Week 12; Part 2: Pre-infusion on Weeks 12, 14, 16, 18, 20, 22, Months 12, 24, 36
Pharmacokinetics of VAL-1221 in Plasma: Terminal Elimination Half-Life ( t1/2) | Part 1: Pre-infusion, end of infusion (EOI) (infusion duration 1 mg/kg/hour), at 0.25, 0.5, 1, 2, 4, 12, 24, 48 and 336 hours after EOI on Days 1, 2, 3 and Week 12; Part 2: Pre-infusion on Weeks 12, 14, 16, 18, 20, 22, Months 12, 24, 36
Pharmacokinetics of VAL-1221 in Plasma: Apparent Total Body Clearance (CL) | Part 1: Pre-infusion, end of infusion (EOI) (infusion duration 1 mg/kg/hour), at 0.25, 0.5, 1, 2, 4, 12, 24, 48 and 336 hours after EOI on Days 1, 2, 3 and Week 12; Part 2: Pre-infusion on Weeks 12, 14, 16, 18, 20, 22, Months 12, 24, 36
Pharmacokinetics of VAL-1221 in Plasma: Apparent Volume (V) | Part 1: Pre-infusion, end of infusion (EOI) (infusion duration 1 mg/kg/hour), at 0.25, 0.5, 1, 2, 4, 12, 24, 48 and 336 hours after EOI on Days 1, 2, 3 and Week 12; Part 2: Pre-infusion on Weeks 12, 14, 16, 18, 20, 22, Months 12, 24, 36
Change from Baseline in Urinary Hexose Tetrasaccharide (hex4) Excretion at Week 12, Months 6, 9, and 12 | Baseline of Study Part 1, Week 12 of Study Part 1, Months 12, 24, and 36 of Study Part 2
Change from Baseline in Serum Creatine Kinase (CK) at Week 12, Months 6, 9, and 12 | Baseline of Study Part 1, Week 12 of Study Part 1, Months 12, 24, and 36 of Study Part 2
Change from Baseline in the Amount of Acid Alpha Glucosidase (GAA) Activity Present in Muscle at Week 12 | Baseline of Study Part 1, Week 12 of Study Part 1
Change from Baseline in the Muscle Glycogen Content at Week 12 | Baseline of Study Part 1, Week 12 Study Part 1
Change from Baseline in Creatinine Excretion at Months 6, 9, and 12 | Baseline of Study Part 1, Months 12, 24, 36 of Study Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Hal Landy, MD, Study Director — Valerion Therapeutics, LLC
Locations (3):
- United States (2):
  - University of California, Irvine, Orange, California
  - Duke University Medical Center, Durham, North Carolina
- National Hospital for Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No